CLINICAL TRIAL: NCT00584064
Title: Emergency/Compassionate Use PFO Occluder
Status: Approved for marketing | Type: Expanded Access
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: AGA-006 - E/C
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Patent Foramen Ovale; PFO
Keywords: patent; foramen; ovale; PFO
MeSH Terms: conditions — Foramen Ovale, Patent

INTERVENTIONS:
Device: Device closure with the AMPLATZER PFO Occluder — Device closure with the AMPLATZER PFO Occluder

SUMMARY:
Emergency/compassionate use for the AMPLATZER PFO Occluder

ELIGIBILITY:
Inclusion Criteria:

* Emergency/compassionate use for patients not meeting the inclusion criteria for the AMPLATZER PFO Access Registry.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult